CLINICAL TRIAL: NCT06866054
Title: Evaluation of the Effectiveness of Ultrasound-Guided Serratus Posterior Superior Intercostal Plane Block for Postoperative Analgesia Management in Patients Undergoing Arthroscopic Shoulder Surgery
Brief Title: Serratus Posterior Superior Intercostal Plane Block for Arthroscopic Shoulder Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Bora Bilal, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-744
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Pain; Shoulder Injuries
Keywords: Arthroscopic Shoulder Surgery; Postoperative analgesia management; serratus posterior superior intercostal plane block
MeSH Terms: conditions — Shoulder Pain; Shoulder Injuries

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is the serratus posterior superior intercostal plane block group. The second one is the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SPSIPB = SPSIPB group (Active Comparator): SPSIPB will be performed
  Interventions: Drug: SPSIPB block; Drug: Postoperative analgesia management
- Group Control (Other): Conventional analgesia management will be performed
  Interventions: Drug: Postoperative analgesia management

INTERVENTIONS:
Drug: SPSIPB block — A high-frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. The procedure will be performed with the patient in the lateral decubitus position. After the scapula is shifted slightly laterally, the US probe is placed sagittal at the upper corner of the spina scapula, and the serratus posterior superior muscle is visualized with the third rib. The in-plane technique will be used. The block needle will be advanced in the craniocaudal direction to enter between the serratus posterior superior and the third rib. The block location will be confirmed by injecting 5 ml of saline between the rib and the muscle. After the block location is confirmed, 30 ml of 0.25% concentration bupivacaine will be used.
  Arms: Group SPSIPB = SPSIPB group
Drug: Postoperative analgesia management — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient-controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol including 10 mcg bolus without infusion dose, 10 min lockout time, and 4-hour limit. If the NRS score is ≥ 4, 0.5 mg kg-1 iv meperidine will be administered as a rescue analgesic. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.

SUMMARY:
Postoperative pain is a significant problem in patients undergoing arthroscopic shoulder surgery. This situation disrupts the patient's comfort and affects the functional outcome after surgery by preventing early rehabilitation. Various methods are used for postoperative pain control. Intravenous opioid agents are one of the most commonly used analgesic techniques. However, opioids can cause undesirable side effects such as respiratory depression, sedation, constipation, allergic reactions, nausea, and vomiting. Therefore, alternative techniques are needed to reduce opioid use.

Serratus posterior superior interfascial plane block (SPSIPB) is a novel interfascial plane block described by Tulgar et al in 2023. It is based on injection into the serratus posterior superior muscle at the level of the 2nd or 3rd rib. This block provides analgesia in cases such as interscapular pain, chronic myofascial pain syndromes, scapulocostal syndrome, and shoulder pain. It has been reported that SPSIPB provides effective shoulder analgesia.

DETAILED DESCRIPTION:
Postoperative pain is a significant problem in patients undergoing arthroscopic shoulder surgery. This situation disrupts the patient's comfort, prevents early rehabilitation, and affects the functional outcome after surgery. Various methods are used for postoperative pain control. Intravenous opioid agents are one of the most commonly used analgesic techniques. However, opioids can cause undesirable side effects such as respiratory depression, sedation, constipation, allergic reactions, nausea, and vomiting. Therefore, alternative techniques are needed to reduce opioid use. Regional techniques can be used for postoperative pain treatment following arthroscopic shoulder surgery. Ultrasound (US)-guided serratus posterior superior block (SPSIPB) is a novel interfascial plane block described by Tulgar et al in 2023. It is based on the principle of injection into the serratus posterior superior muscle at the level of the 2nd or 3rd rib. This block provides analgesia in cases such as interscapular pain, chronic myofascial pain syndromes, scapulocostal syndrome, and shoulder pain. The SPS muscle is located at the C7-T2 level. It attaches to the lateral edges of the second and fifth ribs. It is innervated by the lower cervical and upper intercostal nerves. Analgesia is provided by blocking these nerves with the SPS block. Tulgar et al. reported in their cadaver study that the spread of the serratus posterior superior interfascial plane block; staining in the superficial fascia of the trapezius muscle was observed only on the left side at the 7-10th intercostal levels, but not on the right. There was significant staining deep in the trapezius muscle on both sides. Both the surface and the skin of the rhomboid major were clearly stained, while only the skin of the rhomboid minor was stained; SPSP block will provide successful analgesia in procedures involving the thoracic region such as breast surgery, thoracic surgery, and shoulder surgery.

In this study, the investigators aim to evaluate the analgesic efficacy of SPSIPB by comparing the control group in patients who underwent arthroscopic shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for arthroscopic shoulder surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* patients who do not accept the procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption (Fentanyl PCA) | Changes from baseline opioid consumption at postoperative 1, 2, 4, 8, 16 and 24 hours.
  The primary aim is to compare postoperative opioid consumption from the PCA device.

SECONDARY OUTCOMES:
Pain scores (Numerical rating scale-NRS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16 and 24 hours
  The secondary aim is to compare NRS at the postoperative 24 h. Postoperative pain assessment will be performed using the NRS (0 = no pain, 10 = the most severe pain felt). The NRS scores will be recorded
Need for rescue analgesia (meperidine) | Postoperative 24 hours period
  The secondary aim is to compare rescue analgesia used in the postoperative 24 h.
Adverse events | Postoperative 24 hours period
  The secondary aim is to compare the adverse events (nausea, vomiting, itching) related to opioid use

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medipol University, Istanbul, Bagcilar
  - KSU Faculty of Medicine Research Hospital, Kahramanmaraş

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093
- [Background] Ciftci B, Alver S, Ahiskalioglu A, Bilal B, Tulgar S. Serratus posterior superior intercostal plane block: novel thoracic paraspinal block for thoracoscopic and shoulder surgery. Minerva Anestesiol. 2024 Apr;90(4):345-347. doi: 10.23736/S0375-9393.23.17827-8. Epub 2024 Jan 19. No abstract available. PMID 38240640
- [Background] Ciftci B, Alver S, Ahiskalioglu A, Bilal B, Tulgar S. Serratus posterior superior intercostal plane block for breast surgery: a report of three cases, novel block and new indication. Minerva Anestesiol. 2023 Nov;89(11):1054-1056. doi: 10.23736/S0375-9393.23.17432-3. Epub 2023 Jun 1. No abstract available. PMID 37272274
- [Background] Kulturoglu G, Altinsoy S, Ozguner Y, Cataroglu CK. Novel Serratus Posterior Superior Intercostal Plane Block Provided Satisfactory Analgesia after Breast Cancer Surgery: Two Case Reports. Turk J Anaesthesiol Reanim. 2024 Feb 28;52(1):33-35. doi: 10.4274/TJAR.2024.231431. PMID 38414179
- [Background] Turan EI, Isik S, Baydemir AE, Sahin AS. Serratus posterior superior intercostal plane block for postoperative analgesia in clavicle surgeries: new indications for a novel block. Minerva Anestesiol. 2024 Nov;90(11):1058-1060. doi: 10.23736/S0375-9393.24.18275-2. Epub 2024 Aug 5. No abstract available. PMID 39101308